CLINICAL TRIAL: NCT00318669
Title: Clinical Evaluation of BRL29060A (Paroxetine Hydrochloride Hydrate) in Social Phobia/Social Anxiety Disorder (SAD) -A Double-blind, Placebo-controlled Study- <Phase III Study>
Brief Title: Social Anxiety Disorder Study Of Paroxetine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIR104776
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2012-07

CONDITIONS: Social Phobia
Keywords: Anxiety; SAD; Social; Disorder
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paroxetine hydrochloride hydrate

SUMMARY:
This study is designed to evaluate the efficacy and safety in Social Anxiety Disorder (SAD).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Social Anxiety Disorder (SAD) (300.23 Social Phobia/Social Anxiety Disorder) according to DSM-IV-TR criteria.
* Must give a written informed consent. But if the patient is under 20, both the patient himself/herself and his/her proxy consenter must give written informed consent.
* Patients have a minimum score of 60 on the LSAS total score.

Exclusion criteria:

* Patients primarily diagnosed with a disorder that is categorized into Axis I excluding SAD by DSM-IV-TR (e.g. major depression, dysthymic disorder, specific phobia (simple phobia) , obsessive compulsive disorder, panic disorder) within 24weeks before week -2.
* Patients with a history or complication of schizophrenia and bipolar disorder
* Patients with a complication of body dysmorphic disorder.
* Patients with evidence of substance abuse (alcohol or drugs)
* substance dependence by DSM-IV-TR criteria within 24 weeks before week -2.
* Patients who started psychotherapy and cognitive-behavioural therapy within 24 weeks before week-2, except for supportive psychotherapy.
* Patients receiving electro-convulsive therapy (ECT) within 12 weeks before week -2.
* Patients being pregnant, lactating or are of childbearing potential and are likely to become pregnant.
* Patients with 3 or more points of HAM-D Item No. 3, or who are likely to attempt suicide.
* Patients with a history or complication of cancer or malignant tumor.
* Patients receiving MAO inhibitors (FP®) within 14 days before expected week 0 visit date.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2005-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the LSAS total score at week 12 (Score at week 12 - Score at week 0) | 12 Weeks

SECONDARY OUTCOMES:
Proportion of patients responding with a CGI Global Improvement Item score. Change from baseline in the CGI Severity of Illness score. Change from baseline in the HAM-D total score. Proportion of patients continuing treatment. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site